CLINICAL TRIAL: NCT07397559
Title: Spatiotemporal Control of Transcutaneous Spinal Cord Stimulation for Motor Function in SCI
Brief Title: Spatiotemporal tSCS in Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Ismael Seáñez, Assistant Professor of Biomedical Engineering and Neurosurgery, Washington University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 202506064
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Spinal Cord Injuries (SCI)
Keywords: spinal cord injury; transcutaneous spinal cord stimulation; rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- No stimulation (Other): Participants complete the study motor tasks and assessments without transcutaneous spinal cord stimulation (tSCS).
  Interventions: Other: No Stimulation
- Conventional tSCS (Active Comparator): Participants complete the same experimental tasks and assessments while receiving conventional, non-invasive transcutaneous spinal cord stimulation (tSCS) using a single cathode and 30 Hz.
  Interventions: Device: Conventional tSCS
- Spatiotemporal tSCS (Experimental): Participants complete the same tasks and assessments while receiving spatiotemporal tSCS in which stimulation parameters are systematically varied across sessions, including electrode location/configuration (spatial control), frequency, and amplitude (temporal/intensity control), to optimize targeted muscle recruitment and voluntary motor output.
  Interventions: Device: Spatiotemporal tSCS

INTERVENTIONS:
Other: No Stimulation — Participants complete motor tasks and outcome assessments with no spinal cord stimulation applied.
  Arms: No stimulation
Device: Conventional tSCS — Non-invasive transcutaneous spinal cord stimulation (tSCS) is delivered at 30 Hz using a single cathode electrode targeting the lumbar spinal cord to reinforce leg motor output during study tasks
  Arms: Conventional tSCS
Device: Spatiotemporal tSCS — Stimulation parameters, including electrode location, stimulation frequency, and stimulation amplitude, are systematically varied to reinforce leg motor output during study tasks
  Arms: Spatiotemporal tSCS

SUMMARY:
Spinal cord injury leads to long-lasting impairment, and currently, there is no cure for paralysis. Although transcutaneous spinal cord stimulation has shown promising results in recovering lost movements, its poor selectivity in muscle recruitment compared to invasive approaches limits the type of rehabilitation exercises that can be practiced. This project studies how spatial, frequency, and amplitude control of stimulation can be used to selectively target different neural pathways and muscle groups.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) is a life-altering event that leads to long-lasting motor impairment. Currently, there is no cure for paralysis. Transcutaneous spinal cord stimulation (tSCS) combined with exercise training can restore posture control, voluntary walking, and arm/hand function in people with SCI. However, its low selectivity in activating specific muscles compared to invasive approaches limits the rehabilitation exercises that can be practiced and help with recovery. This project will generate evidence-based knowledge of the neural mechanisms underlying spatial, frequency, and amplitude control of tSCS in generating different types of leg movements. Participants with SCI will perform leg movements using different stimulation parameter configurations in non-invasive tSCS. We will quantify changes in muscle recruitment, torque generation, and pain enabled by the different stimulation parameters. A clear understanding of the mechanisms by which these different parameters in non-invasive tSCS can be used to selectively target different muscle groups will promote the development of personalized therapies that directly target only those muscles that need assistance while respecting individuals' residual motor function.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 16 and 65 years.
2. Have a spinal cord injury (neurological level C3-T12) that occurred ≥1 year (chronic stage) prior to enrollment.
3. American Spinal Injury Association (ASIA) Impairment Scale (AIS) classification C or D
4. Able to voluntarily contract (motor score ≥ 1) at least two leg muscles (visual or palpable contraction).
5. Use of prescription medication(s) for control of spasticity has not changed in the last 2 weeks
6. Able to provide consent
7. Ability to follow multiple instructions and communicate pain or discomfort

Exclusion Criteria:

1. Progressive spinal lesions, including degenerative disorders of the spinal cord
2. Pregnant, planning to become pregnant, or currently breastfeeding
3. History of cardiopulmonary disease or cardiac symptoms
4. Implanted stimulators of any type (baclofen pump, epidural spinal stimulator, cardiac defibrillator, pace-maker, etc.)
5. Presence of orthopedic conditions that would negatively affect participation in leg exercise
6. History of autonomic dysreflexia that is severe, unstable, and/or uncontrolled
7. Unstable or significant medical conditions that can interfere with exercise or neurophysiological evaluations, such as severe neuropathic pain, depression, mood disorders, or other cognitive disorders
8. Spasms that limit the ability to participate in leg exercise activity
9. Breakdown in skin area that will be in contact with electrodes

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-01-19 (Actual); Primary Completion 2030-08-31 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Torque | 30 minutes
  The primary outcome is a measure of changes in voluntary torque production (Nm)

SECONDARY OUTCOMES:
Muscle activation | 30 minutes
  Muscle activation will be measured through electromyography as the peak-to-peak of the evoked responses (mV)
Pain/Nociception | 30 minutes
  Pain will be evaluated using the Nociception Level (NOL) index during the different stimulation conditions. (Range: 0-100, 0 = no detectable nociceptive response, 100 = extreme nociceptive response)

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University, St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified and anonymized individual participant data including kinematic measures, EMG torque, stimulation parameters, nociception/pain measures, and associated session/task metadata. Processed datasets and summary statistics used for publications will be shared. Identifiable video recordings will not be shared.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: IPD and supporting information will be made available no later than the time of publication of the primary results and/or at the end of the study performance period, whichever occurs first. Data will remain available for at least 5 years following the end of the study, subject to repository policies and continued availability of the hosting platforms.
Access Criteria: Access will be provided to qualified researchers for non-commercial scientific purposes. Shared datasets will be de-identified/anonymized and will not include direct identifiers or any information that could reasonably be used to re-identify participants. Data will be accessed via public repositories when available (e.g., Open Data Commons for Spinal Cord Injury) and/or through controlled-access request mechanisms (e.g., NICHD DASH) as applicable.
URL: https://seanezlab.wustl.edu/data-sharing/